CLINICAL TRIAL: NCT02614586
Title: A Placebo-Controlled Study to Evaluate the Effect of a Single Dose of TAK-058 and Ondansetron on P50 Auditory Gating in Subjects With Stable Schizophrenia
Brief Title: Evaluation of TAK-058 and Ondansetron on P50 Auditory Gating in Participants With Stable Schizophrenia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-058-1003; U1111-1168-1522 (Registry Identifier: WHO)
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia
Keywords: Drug Therapy
MeSH Terms: conditions — Schizophrenia | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo + TAK-058 + Ondansetron (Experimental): TAK-058 placebo-matching solution, orally, along with ondansetron placebo-matching capsule, orally, on Day 1 of first intervention period (2 days), followed by 1 week washout period, further followed by TAK-058 150 milligram (mg), solution, orally along with ondansetron placebo-matching capsule orally, on Day 1 of second intervention period (2 days), followed by 1 week washout period, further followed by ondansetron 16 mg, capsule, orally along with TAK-058 placebo-matching solution, orally, on Day 1 of third intervention period (2 days).
  Interventions: Drug: TAK-058; Drug: Ondansetron; Drug: TAK-058 Placebo; Drug: Ondansetron Placebo
- TAK-058 + Placebo + Ondansetron (Experimental): TAK-058 150 mg, solution, orally along with ondansetron placebo-matching capsule orally, on Day 1 of first intervention period (2 days), followed by 1 week washout period, further followed by TAK-058 placebo-matching solution, orally, along with ondansetron placebo-matching capsule, orally, on Day 1 of second intervention period (2 days), followed by 1 week washout period, further followed by ondansetron 16 mg, capsule, orally, along with TAK-058 placebo-matching solution, orally, on Day 1 of third intervention period (2 days).
  Interventions: Drug: TAK-058; Drug: Ondansetron; Drug: TAK-058 Placebo; Drug: Ondansetron Placebo
- Ondansetron + Placebo + TAK-058 (Experimental): Ondansetron 16 mg, capsule, orally, along with TAK-058 placebo-matching solution, orally, on Day 1 of first intervention period (2 days), followed by 1 week washout period, further followed by TAK-058 placebo-matching solution, orally, along with ondansetron placebo-matching capsule, orally, on Day 1 of second intervention period (2 days), followed by 1 week washout period, further followed by TAK-058 150 mg, solution, orally, along with ondansetron placebo-matching capsule, orally, on Day 1 of third intervention period (2 days).
  Interventions: Drug: TAK-058; Drug: Ondansetron; Drug: TAK-058 Placebo; Drug: Ondansetron Placebo
- Placebo + Ondansetron + TAK-058 (Experimental): TAK-058 placebo-matching solution, orally, along with ondansetron placebo-matching capsule, orally, on Day 1 of first intervention period (2 days), followed by 1 week washout period, further followed by ondansetron 16 mg, capsule, orally, along with TAK-058 placebo-matching solution, orally, on Day 1 of second intervention period (2 days), followed by 1 week washout period, further followed by TAK-058 150 mg, solution, orally, along with ondansetron placebo-matching capsule, orally, on Day 1 of third intervention period (2 days).
  Interventions: Drug: TAK-058; Drug: Ondansetron; Drug: TAK-058 Placebo; Drug: Ondansetron Placebo
- TAK-058 + Ondansetron + Placebo (Experimental): TAK-058 150 mg, solution, orally along with ondansetron placebo-matching capsule orally, on Day 1 of first intervention period (2 days), followed by 1 week washout period, further followed by ondansetron 16 mg, capsule, orally, along with TAK-058 placebo-matching solution, orally, on Day 1 of second intervention period (2 days), followed by 1 week washout period, further followed by TAK-058 placebo-matching solution, orally, along with ondansetron placebo-matching capsule, orally, on Day 1 of third intervention period (2 days).
  Interventions: Drug: TAK-058; Drug: Ondansetron; Drug: TAK-058 Placebo; Drug: Ondansetron Placebo
- Ondansetron + TAK-058 + Placebo (Experimental): Ondansetron 16 mg, capsule, orally along with TAK-058 placebo-matching solution, orally, on Day 1 of first intervention period (2 days), followed by 1 week washout period, further followed by TAK-058 150 mg, solution, orally, along with ondansetron placebo-matching capsule, orally, on Day 1 of second intervention period (2 days), followed by 1 week washout period, further followed by TAK-058 placebo-matching solution, orally, along with ondansetron placebo-matching capsule, orally, on Day 1 of third intervention period (2 days).
  Interventions: Drug: TAK-058; Drug: Ondansetron; Drug: TAK-058 Placebo; Drug: Ondansetron Placebo

INTERVENTIONS:
Drug: TAK-058 — TAK-058 oral solution.
Drug: Ondansetron — Ondansetron capsule.
Drug: TAK-058 Placebo — TAK-058 placebo-matching, solution.
Drug: Ondansetron Placebo — Ondansetron placebo-matching, capsule.

SUMMARY:
The purpose of this study is to determine whether improvement in P50 (a pharmacodynamic marker) in auditory sensory gating is demonstrated after administration of TAK-058 and ondansetron compared to placebo in participants with schizophrenia.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-058. TAK-058 is being tested to evaluate its effects on P50 auditory gating in people who have stable schizophrenia. This study will look at the effect of TAK-058 on P50 auditory gaiting of people with schizophrenia.

This study will be performed in a sequential manner progressing from an optimization (screening) phase in healthy volunteers, to screening of subjects with schizophrenia in part 1, to a 3 period crossover treatment phase in part 2. In the screening phase, 15 healthy volunteers will be enrolled to optimize the settings for the measurement of neurophysiological markers prior to any dosing in participants with schizophrenia. If optimization is not reached, the study will be terminated. In part 1 participants with schizophrenia will receive 2 P50 electroencephalography (EEG) sessions. A measurable deficit in auditory P50 gating S2/S1 ratio greater than (>) 0.5 will be established during this phase. The intraclass correlation coefficient (ICC) will be calculated for the P50 auditory gating S2/S1 ratios collected during the 2 sessions. If these P50 auditory gating S2/S1 ratio measurements are found to have at least a fair level of agreement within individuals (that is, ICC > 0.5), part 2 of the study will begin. 12 participants demonstrating P50 impairment in part 1, will be randomly assigned (by chance, like flipping a coin) to one of the six treatment crossover sequences -which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Placebo + TAK-058 + Ondansetron
* TAK-058 + Placebo + Ondansetron
* Ondansetron + Placebo + TAK-058
* Placebo + Ondansetron + TAK-058
* TAK-058 + Ondansetron + Placebo
* Ondansetron + TAK-058 + Placebo

All participants will be asked to take one dose of capsule, followed 1 hour later by one dose of solution on Day 1 of each intervention period.

This single-center trial will be conducted in the United States. The overall time to participate in this study is approximately 118 days. Participants will make be confined to the clinic for 3 days (Day -1 through Day 2 of each period), a final visit for schizophrenic participants in Part 2 after receiving TAK-058, on Day 2 of Period 3 (no final visit for optimization phase healthy participants), and a telephonic follow up assessment 21 days after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 60 years of healthy and schizophrenic participants, inclusive, at the time of informed consent.
2. Has acceptable clinical laboratory evaluations (including clinical chemistry, hematology and complete urinalysis).
3. Meets schizophrenia criteria as defined by the Diagnostic & Statistical Manual of Mental Disorders, 5th Edition (DSM-V).
4. Are on a stable dose of single second-generation antipsychotics (SGA) for at least 2 months prior to Screening as documented by medical history and assessed by site staff.
5. Demonstrates Positive and Negative Syndrome Scale (PANSS) total score of less than equal to (<=) 85.
6. Has a P50 ratio of > 0.5 at both screening assessments.

Exclusion Criteria:

1. Has a history in the last year or currently receiving treatment with clozapine or olanzapine.
2. Has taken any excluded medications, supplements or food products.
3. Has a history of gastrointestinal disease that would influence the absorption of study drug or have a significant medical history of any disease that would contraindicate the administration of TAK-058, ondansetron, or a similar compound.
4. Has substance abuse or dependence within previous 12 months, unstable mood or anxiety disorder.
5. Has a current diagnosis of a significant psychiatric illness other than schizophrenia per DSM-V and is in an acute phase/episode.
6. Has clinically meaningful hearing loss per investigator's judgment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 09 December 2015 to 29 April 2016.
Pre-assignment Details: Participants with a diagnosis of schizophrenia were enrolled in this 2-part study comprised of Part-1, screening and Part-2, treatment phase. Part-2 was not initiated because in Part-1 (sequential step 2), the P50 auditory gating (stimulus[S]2/S1) ratio for alpha and beta frequency bands demonstrated high variability and the study was terminated.
Groups:
- Part-1: Screening Phase: Participants received 2 P50 electroencephalography (EEG) sessions, first session was conducted in the morning, and second session was conducted in the afternoon. Participants did not receive any study medication in Screening Phase (Part-1) of the study.
Period: Overall Study
Arm/Group | Part-1: Screening Phase
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Schizophrenia Set included all participants who were enrolled and completed the Screening Phase (Part-1) of the study.
Arm/Group | Part-1: Screening Phase
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (4.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 11
Region of Enrollment [Number; unit: participants]
  United States | 11
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 170.7 (12.39)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 87.75 (19.351)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 29.93 (4.929)
Smoking Classification [Number; unit: participants]
  Never Smoked | 6
  Current Smoker | 5
Caffeine Consumption [Number; unit: participants]
  Consumed Caffeine | 9
  Did not Consume Caffeine | 2
Female Reproductive Status [Number; unit: participants] — Reproductive status was not applicable for male participants.
  participants
    Postmenopausal | 1
    Surgically Sterile | 1
    Have Childbearing Potential | 3
    Not Applicable | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in P50 Ratio S2/S1 at Central (Cz) Electrode Following Administration of TAK-058
Description: Participants were planned to check for P50 gating ratio. Stimulus signal of 90 decibel pulses of 0.1 millisecond (msec) was to be generated and recorded the event-related potential waveforms. 32 pairs of auditory clicks were to be presented every 10 seconds, with a 500 msec interclick interval. S1 is defined as the conditioning P50 wave with the most positive peak between 30 and 90 msec after the conditioning stimulus. S2 is defined as the test P50 wave with the positive peak after the test stimulus that was closest in latency to the conditioning P50. Amplitude is the difference between the positive peak and the preceding negative trough for both waves. The data from the vertex (Cz site) was to be collected and the P50 gating ratio (S2/S1) was to be calculated as the ratio of the test P50 amplitude to the conditioning P50 amplitude.
Time Frame: Part 2: Day 1 pre-dose and at multiple time points (up to 2 hours) post-dose in each period.
Population: Part 2 was not initiated because it was not possible to calculate an ICC due to the magnitude of the intrasubject variability in relation to the intersubject variability.
Groups:
- Part 2: TAK-058 and Ondansetron: In Treatment Phase (Part 2) of the study, participants were planned to be randomized into 3-period cross-over treatment phase with single oral dose of 1 of the 3 regimens in each period: TAK-058, ondansetron, and placebo. Participants were planned to receive treatment in following 6 sequences: placebo, TAK-058, and ondansetron; TAK-058, placebo, and ondansetron; ondansetron, placebo, and TAK-058; placebo, ondansetron, and TAK-058; TAK-058, ondansetron, and placebo; and ondansetron, TAK-058, and placebo in intervention period 1, 2, and 3 respectively. A washout period of at least 7 days was planned to be maintained between each intervention period.
Arm/Group | Part 2: TAK-058 and Ondansetron
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Time Frame: Part 2: Day 1 of Intervention Period 1 up to Day 21
Population: as for outcome 1
Arm/Group | Part 2: TAK-058 and Ondansetron
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 of Period 1 of Part 2, up to 21 days after last dose of study drug in Part 2
Description: No AE assessments were done because AEs were planned to be collected in Treatment Phase (Part-2) of the study which was not initiated because it was not possible to calculate an ICC due to the magnitude of the intrasubject variability in relation to the intersubject variability.
Arm/Group | Part 2: TAK-058 and Ondansetron
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.